CLINICAL TRIAL: NCT00913679
Title: A Comparison of Two Different Surgical Techniques to Preserve the Bony Supply and Improve Implant Longevity in Hip Resurfacing Arthroplasty
Brief Title: A Comparison of Two Different Surgical Techniques in Hip Resurfacing Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20070082
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Osteonecrosis; Femoral Neck Fracture; Implant Failure
Keywords: osteonecrosis; femoral neck fracture; implant fixation; implant failure; periprosthetic bone mineral density; gait function; gait analysis; patient recovery
MeSH Terms: conditions — Osteonecrosis; Femoral Neck Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Posterior approach (Active Comparator): Posterior surgical approach in hip resurfacing arthroplasty
  Interventions: Procedure: Surgical approach (ReCap Hip Resurfacing System)
- Anterolateral approach (Active Comparator): Anterolateral surgical approach in hip resurfacing arthroplasty
  Interventions: Procedure: Surgical approach (ReCap Hip Resurfacing System)

INTERVENTIONS:
Procedure: Surgical approach (ReCap Hip Resurfacing System) — two different surgical approaches in hip resurfacing arthroplasty
  Other Names: ReCap Hip Resurfacing System

SUMMARY:
The purpose of the study is to compare two different surgical techniques in hip resurfacing arthroplasty (RHA), comparing bloodflow and metabolism in the femoral head, as well as implant migration, periprosthetic bone mineral density, gait function and patient recovery.

DETAILED DESCRIPTION:
BACKGROUND:

6700 total hip replacements are performed each year in Denmark due to osteoarthritis. Young patients sustain a substantial risk of early implant failure due to high-activity daily living, and among patients younger than 55 years at surgery 20 percent need revision surgery within ten years. Revision surgery is more complicated than primary surgery and associated with decreased implant longevity due to decreased bone stock. Resurfacing hip arthroplasty (RHA), restores the anatomy of the hip as only the articulating joint surfaces are replaced, and thus more bone is left to ensure a better opportunity of successful revision surgery later on. The clinical midterm evaluation of RHA survival is promising, but two major complications leading to early revision, namely osteonecrosis and femoral neck fracture, has raised concern regarding the influence of surgical technique on the vascularity of the femoral head. RHA is commonly performed through a posterolateral surgical approach. By this technique muscle tendons are spilt resulting in decreased patient mobility for several weeks after surgery, but more importantly, the blood supply is compromised as a large artery has to be ligated. This is speculated to decrease the blood supply to femoral head and neck and thereby increase the risk of osteonecrosis, femoral neck fracture, and implant failure. With a new surgical technique facilitating an anterolateral approach to the hip joint the blood supply is left intact as well as the muscle tendons.

HYPOTHESIS:

An anterolateral surgical approach in resurfacing hip arthroplasty will 1) preserve the blood supply to the femoral head and neck and improve implant longevity, and 2) spare the muscle tendons and ease patient recovery.

METHOD and FACILITIES:

50 patients, aged 30 to 60 years, with osteoarthrosis of the hip will be randomised to a RHA inserted by either an anterolateral or a posterolateral surgical approach. Primary points of evaluation are 1) blood supply to the femoral head and neck measured intraoperatively by Laser Doppler flowmetry and postoperatively by microdialysis established during surgery. Secondary points of evaluation are 1) implant fixation measured by radiostereometric analysis (RSA), and 2) periprosthetic bone mineral density (BMD) measured by dual energy x-ray absorptiometry (DEXA), 3) gait analysis and 4) clinical scores of function, pain and activities of daily living (Harris Hip Score , Visual Analogue Scale).

ELIGIBILITY:
Inclusion Criteria:

* Primary hip OA;
* Secondary hip OA due to mild and moderate acetabular dysplasia;
* Sufficient bone quality for cementless acetabular component;
* Suited for resurfacing of the femoral head, pre and intraoperatively assessed;
* Age 30 to 60 years.

Exclusion Criteria:

* Neuromuscular or vascular diseases in affected leg;
* Patients found intra-operatively to be unsuited for a cementless acetabular component or cementing of the femoral component;
* Need of NSAID postoperatively;
* Fracture sequelae;
* Females at risk of pregnancy, no safe contraceptives;
* Severe hip dysplasia;
* Sequelae from hip disease in childhood;
* Medicine with large effect on bone density, K vitamin antagonists, loop-diuretics;
* Alcoholism, females over 14 units per week, males over 21 units per week; AVN;
* Osteoporosis.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2008-11-01 (Actual); Primary Completion 2017-02-20 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
femoral head blood flow, evaluated by Laser Doppler Flowmetry | during surgery
femoral head metabolism, evaluated by microdialysis | 3 days

SECONDARY OUTCOMES:
implant fixation, evaluated by RSA (radiostereogrammetric analysis) | postoperatively; 3 months; 1,2 and 5 years
periprosthetic bone mineral density, evaluated by DEXA | pre- and postoperatively; 1 and 2 years
gait function, evaluated by gait analysis | preoperatively; 3 months and 1 year
patient recovery, evaluated by Harris Hip Score and Visual Analogue Scale | preoperatively and 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Department of Orthopaedic Surgery, Tage-Hansens Gade 2, Aarhus C, Aarhus County, Denmark

REFERENCES:
- [Derived] Jorgensen PB, Krag-Nielsen N, Lindgren L, Morup RMS, Kaptein B, Stilling M. Radiostereometric analysis: comparison of radiation dose and precision in digital and computed radiography. Arch Orthop Trauma Surg. 2023 Sep;143(9):5919-5926. doi: 10.1007/s00402-022-04674-0. Epub 2022 Nov 23. PMID 36422666